CLINICAL TRIAL: NCT01552044
Title: Evaluation de la Spironolactone Dans le Traitement Des choriorétinites séreuses Centrales Non résolutives à Trois Mois
Brief Title: Effect of Spironolactone in Treating Chronic Non-resolutive Central Serous Chorioretinitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C11-21; 2011-003046-40 (EudraCT Number)
Record Dates: First submitted 2012-02-14; First posted 2012-03-13 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2016-02

CONDITIONS: Central Serous Chorioretinitis
Keywords: retina
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- spironolactone (Experimental): Spironolactone 25mg/day
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25mg tablet once a day for 1 month
  Other Names: aldactone
  Arms: spironolactone
Drug: Placebo — one tablet once a day for 1 month
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the effect of spironolactone on 16 patients presenting with chronic non-resolutive central serous chorioretinitis (CSCR) and to evaluate whether spironolactone can resolve sub retinal fluid in these patients.

CSCR is a major cause of visual loss in the young population. It is characterized by sub retinal fluid under the retina and retinal pigment epithelial detachments. The exact causes of the disease remain unknown but a choroidopathy has been suggested. Moreover, corticotherapy and stress are known risk factors of CSCR.

Our preclinical studies have demonstrated that the mineralocorticoid pathway could be involved in the control of choroidal blood flow.

The investigators propose to evaluate the mineralocorticoid receptors antagonist spironolactone in the treatment of CSCR.

Criteria of efficacy Endpoint: reduction of subretinal fluid ≥ 40 microns Secondary endpoint: visual acuity gain ≥ 15 EDTRS letters

DETAILED DESCRIPTION:
This is a prospective placebo controlled cross over study including 16 patients

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 60 years
* CSCR affecting the macula and non-resolutive for at least 3 months
* Patients having given and signed informed consent
* Vital prognosis non engaged for the next 6 months.

Exclusion Criteria:

* Other ocular pathology
* Neovascularization,
* Diabetes
* Uveitis
* Ocular surgery in the last 3 months
* Allergy to fluorescein or indocyanine green
* Pregnancy or no contraception
* Renal or liver insufficiency
* Kaliemia ≥ 5.5 mmol/l Criteria of efficacy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in Central macular thickness | 1 and 3 months
  Sub retinal fluid decrease > or = 40 microns

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel-Dieu of Paris, Paris, France

REFERENCES:
- [Background] Bousquet E, Beydoun T, Rothschild PR, Bergin C, Zhao M, Batista R, Brandely ML, Couraud B, Farman N, Gaudric A, Chast F, Behar-Cohen F. SPIRONOLACTONE FOR NONRESOLVING CENTRAL SEROUS CHORIORETINOPATHY: A RANDOMIZED CONTROLLED CROSSOVER STUDY. Retina. 2015 Dec;35(12):2505-15. doi: 10.1097/IAE.0000000000000614. PMID 26017871
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203